CLINICAL TRIAL: NCT05443815
Title: Prospective Multicenter Registry on the Use of HaemoCer-PLUSPlus in the Treatment and Prevention of Post-resectional Bleeding
Brief Title: Registry on the Use of HaemoCER-Plus in the Treatment and Prevention of Post-resectional Bleeding
Acronym: HemoCER
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istituto Clinico Humanitas Mater Domini (Other)
Responsible Party: Sponsor
Other Study IDs: 11
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Post-resectional Bleeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HaemoCer-PLUS: Patients who had receive HaemoCer-PLUS
  Interventions: Device: HaemoCer-PLUS

INTERVENTIONS:
Device: HaemoCer-PLUS — HaemoCer-PLUS

SUMMARY:
Gastrointestinal bleeding is defined as clinical evidence of bleeding manifested by melena, hematochezia that required endoscopic hemostasis. GI bleeding associated to endoscopic procedure is defined as clinical evidence of bleeding and a drop in hemoglobin of ≥ 2g/dL on the day of the procedure (early bleeding) or up to 14 days after the procedure (delayed bleeding).GI bleeding is, nevertheless, a common complication of endoscopic procedures, such as endoscopic mucosal resection (EMR) and endoscopic sub mucosal dissection (ESD). For example, colorectal ESD, which is technically more difficult than gastric or esophageal ESD because of the anatomical features of the colon, present an increased risk of delayed bleeding. According to literature, early bleeding occurs on average in 5,3% of endoscopic resections of the whole digestive tract, with bleeding rates per location as follows: esophagus 9.4%, stomach 9.1%, duodenum 3.6%, colon 3.4%. Concerning delayed bleeding, it is assessed to complicate 3.1% of endoscopic resection procedures. The bleeding rate in the duodenum is usually the highest (6.3%), followed by colon at (3.6%), stomach (1.5%) and esophagus (0.9%). Age, lesion size and piecemeal resection are associated with an increased risk of bleeding. Usage of aspirin or NSAIDs seems to not increase risk of post-polypectomy bleeding, while clopidogrel and warfarin do and should be discontinued in the periprocedural period to prevent the occurrence of post-polypectomy bleeding. Direct oral anticoagulants (DOAC) administration shows similar post-procedural gastrointestinal bleeding risk to anti-vitamin K antagonists (VKA) administration in patients undergoing endoscopic procedures.

ELIGIBILITY:
Inclusion Criteria:

* patients who had authorized to use and process their personal details for the purpose of research;
* patients able to express their consent;
* age >18 years;
* endoscopic procedures where HaemoCer-PLUS has been used for hemostasis or prevention of bleeding

Exclusion Criteria:

* hemostatic therapies other than HaemoCer-PLUS
* Known coagulopathy likely to affect risk of bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This will be a multicenter and observational registry of patients treated with HaemoCer- PLUS to obtain hemostasis.
  All centres participating in the project will select the patients according to the in- and exclusion criteria. Ethical approval will be obtained in every participant hospital. All patients entering this new registry will have to sign a patient inform consent.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Number and proportion of bleeding events in patients receiving HaemoCer-PLUS | 6 months
  Number and proportion of bleeding events controlled by application of HaemoCer

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas-Mater Domini, Castellanza, Italy

IPD SHARING:
Plan to Share IPD: No